CLINICAL TRIAL: NCT01674348
Title: A Phase II, Randomized, Double-blind, Placebo-controlled, Dose-ranging, Two-staged, Fixed Design Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of P2202 in Overweight/Obese Patients of Type 2 Diabetes Mellitus Inadequately Controlled on Metformin, Sulphonylurea, or Both.
Brief Title: A Clinical Trial to Study the Efficacy, Safety, Tolerability and Pharmacokinetics of P2202 in Patients of Type 2 Diabetes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to non-recruitment, the study is being halted. There are no major safety or tolerability concerns in the study conducted so far.
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P2202/47/10
Record Dates: First submitted 2012-08-21; First posted 2012-08-28 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- P2202 (Active Comparator): Two treatment arms in Stage I- P2202 (1000 mg) and placebo
  Four treatment arms in stage II- P2202 (suggested dose levels 750 mg, 500 mg or 250 mg) or placebo
  Interventions: Drug: P2202
- Placebo (Placebo Comparator): Two treatment arms in Stage I- P2202 (1000 mg) and placebo
  Four treatment arms in stage II- P2202 (suggested dose levels 750 mg, 500 mg or 250 mg) or placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: P2202 — Novel oral drug with potent and selective 11 beta-hydroxysteroid dehydrogenase type 1 (11b-HSD1) inhibitory properties, being developed for the management of type 2 diabetes mellitus
  Arms: P2202
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
It is a phase II, randomized, double-blind, placebo-controlled study of P2202 in patients of type 2 diabetes mellitus, inadequately controlled with a stable dose of metformin or sulfonylurea or both.

DETAILED DESCRIPTION:
It is a phase II, prospective, randomized, double-blind, placebo-controlled, dose-ranging, multi-centre, two-staged, fixed-design study of P2202 in patients of type 2 diabetes mellitus, inadequately controlled with a stable dose of metformin or sulfonylurea or both. This study will consist of accrual in Stage I (n=56/arm, which is 70% of the total sample size required), followed by an interim analysis on completion of the treatment period, to aid further decisions on accrual and dose selection in Stage II of the study, and completion of Stage I.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who understand and are willing to give informed consent to participate in the trial.
* Adult male and female subjects between 18 years to 65 years of age with a BMI ≥ 27 kg/m2 ≤ 40 kg/m2, inclusively.
* Subjects with established type 2 diabetes mellitus of at least 3 months duration at the time of screening.
* Subjects with an inadequate glycemic control defined by an HbA1c level of ≥ 7.5% and ≥10% at screening.
* Subjects who are on a stable dose of:

  * Metformin (up to 2.55 gm/day or maximum tolerated dose of at least 1 gm/day) and/or
  * Sulfonylurea (glimepiride ≤ 4 mg/day, gliclazide ≤ 160 mg, glibenclamide or glyburide ≤ 10 mg and glipizide ≤ 10 mg), for ≤ 2 months prior to the screening visit.
* Subjects with fasting plasma glucose of ≤14.4 mmol/L (260 mg/dL) and at least 5.5 mmol/L or 100 mg/dL.

Exclusion Criteria:

* Subjects who have type 1 diabetes mellitus, maturity-onset diabetes of the young or any rare form of diabetes. Subjects with hyperglycemia due to secondary causes.
* Subjects who have had more than 4 episodes of severe hypoglycemia in the 6 months prior to screening.
* Subjects with a history of acute diabetic complications
* Subjects who have been treated with insulin (except for use of insulin for short term management of acute conditions), thiazolidinediones, dual proliferator activated receptors agonists, glucagon-like peptide analogues, dipeptidyl peptidase inhibitors or 11bHSD-1 inhibitors in any form, in the 3 months prior to screening.
* Subjects who are receiving systemic glucocorticoids (≥14 days)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline | From baseline till end of 12 weeks
  The change in HbA1c from baseline till end of 12 weeks in patients of type 2 diabetes mellitus, in the P2202 arms as compared to placebo.

SECONDARY OUTCOMES:
Number of subjects with adverse events | From screening to 3 weeks (± 1 week) after the last visit at the end of Week 12 or early exit visit
  Safety assessment will be done by eliciting information regarding AEs including evaluation of hypoglycemic events, physical examination, vital signs assessment, 12-lead ECGs, clinical laboratory tests, markers of HPA axis function, plasma ACTH and free testosterone, plasma rennin and serum aldosterone and self-monitoring of blood glucose profiles.

OTHER OUTCOMES:
Pharmacokinetic profile (Cmax, Tmax and AUC) | Pre dose at Day 1 Week 1 till Week 12
  PK parameters derived will be maximum plasma concentration (Cmax), time at which Cmax is reached (Tmax), area under the plasma concentration curve calculated up to 24 hours (AUC 0-24h), area under the curve extrapolated to infinity (AUC 0-inf), elimination rate constant (Kel), volume of distribution (Vz), terminal elimination half life (t1/2) and protein binding.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ronnie Aronson, M.D., Principal Investigator — Health Canada; Dr. Robert Petrella, M.D., Principal Investigator — Health Canada; Dr. Naresh Aggarwal, M.D., Principal Investigator — Health Canada
Locations (1):
- LMC Endocrinolgy Centres Ltd, Toronto, Ontario, Canada